CLINICAL TRIAL: NCT01465698
Title: Effectiveness and Financial Feasibility of Neuromuscular Exercise and Counselling Interventions on Pain, Movement Dysfunction, and Fear-avoidance Behaviour in Female Nurses With Non-specific Low Back Pain
Brief Title: Prevention of Chronic Low Back Pain in Female Nurses
Acronym: NURSE-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UKK Institute (Other)
Collaborators: Tampere University Hospital (Other); Finnish Institute of Occupational Health (Other); University of Zurich (Other)
Responsible Party: Principal Investigator, Jaana Suni, Senior Reseracher, UKK Institute
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R08157
Record Dates: First submitted 2011-10-28; First posted 2011-11-07 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Low Back Pain
Keywords: exercise; counseling; movement control; fear avoidance
MeSH Terms: conditions — Low Back Pain; Motor Activity | interventions — Exercise; Muscle Stretching Exercises; Physical Fitness; Counseling; Behavior Therapy; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Exercise (Experimental)
  Interventions: Behavioral: Exercise
- Counseling (Experimental)
  Interventions: Behavioral: Counseling
- Exercise and counseling (Experimental)
  Interventions: Behavioral: Exercise and counseling
- Control group (Other): Participants in the control group only participate in study measurements.
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Exercise — The main target for exercise intervention is to restore impairments in movement control. First, the participants need to learn the proper technique of each exercise, second to achieve movement control of lumbar neutral zone in each exercise, and finally to increase the challenge of exercises for balance, coordination, muscular endurance and strength. Target dose for exercise is twice a week, 60 minutes per session for six months.
  The neuromuscular exercise program is progressive including three different performance levels. During the first eight weeks, the supervised exercise sessions will take place twice a week. The next 16 weeks the participants have one instructed weekly session, and they exercise once a week at home with help of a DVD or booklet produced for the study
  Other Names: Neuromuscular exercise; Control of lumbar neutral zone; Physical fitness
  Arms: Exercise
Behavioral: Counseling — Counseling is conducted according cognitive-behavioral principles. Fear-avoidance model is implemented using problem based learning. The objective is to change participants' understanding of LBP towards less fearful and negative beliefs, and to provide encouragement for usual daily activities, including physical activity. Advice on nursing tasks that are strenuous for low back is aimed to improve awareness of injury risk and provide examples of proper postures and movements. The target is that participants in counseling groups attend 10 sessions each lasting 45 minutes. During the first four weeks the groups meet every second week, and after that once a month up to six months. Participants will receive workbooks to enhance problem-based learning.
  Other Names: Behavioral counseling; Fear avoidance beliefs; Physical activity promotion
  Arms: Counseling
Behavioral: Exercise and counseling — Participants take part in both exercise and counseling as described in the separate interventions.
  Other Names: Neuromuscular exercise; Control of lumbar neutral zone; Physical fitness; Behavioral counseling; Fear avoidance beliefs; Physical activity promotion
  Arms: Exercise and counseling
Other: Control group — Participants in the control group take part only in measurements of NURSE-RCT.
  Other Names: No intervention
  Arms: Control group

SUMMARY:
NURSE-RCT is a randomized controlled trial which aims at prevention of evolution of chronic low back pain (LBP) and related disability in female nurses.

The study investigates the effectiveness and financial feasibility of six months neuromuscular training and counselling, and their combination on LBP, movement dysfunction and fear-avoidance behaviour.

The target for neuromuscular training is to reduce movement dysfunction and motor control impairments, caused by trauma and subfailure injuries of spinal ligaments. Training aims at enhancement of motor control of lumbar neutral zone in different positions and movements, balance, coordination, trunk muscle endurance and leg strength.

The target for counselling is change in attitudes and behaviour, which help to reduce the fear of pain and encourage to physical activity and other physical tasks.

The hypothesis is that together neuromuscular exercise and counselling have a stronger influence on LBP, movement dysfunction and fear-avoidance behaviour than either used alone.

Assessments of effectiveness will be conducted after six, 12, and 24 months of the beginning of interventions.

DETAILED DESCRIPTION:
Musculoskeletal disorders are the main reason for work absenteeism and early retirement of nursing stuff, low back pain (LBP) being the leading cause. When compared to other communal staff in Finland, disability pensions are granted earlier to nursing stuff, the average age being 56 years. NURSE-RCT is a multidisciplinary study combining the most recent biomechanical and behavioral theories aimed to prevent evolution of chronic LBP.

NURSE-study is a randomized controlled trial aiming at prevention of chronic LBP and related functional disability. Volunteers, female nurses (n~1200) from wards with bed patients of two geriatric hospitals and the university central hospital in Tampere, Finland will be invited to participate in the study. Each participant (n=160) will be randomized into one of the four study groups after the eligibility has been determined. A method of sequentially numbered sealed envelopes will be used to assign participants into study groups.

The main target for exercise intervention is to restore impairments in movement control. First, the participants need to learn the proper technique of each exercise, second to achieve movement control of lumbar neutral zone in each exercise, and finally to increase the challenge of exercises for balance, coordination, muscular endurance and strength. Target dose for exercise is twice a week, 60 minutes per session for six months.

The objective of counseling is to change participants' understanding of LBP towards less fearful and negative beliefs, and to provide encouragement for usual daily activities, including physical activity. Advice on nursing tasks that are strenuous for low back is aimed to improve awareness of injury risk and provide examples of proper postures and movements. Target dose for counseling is 10 sessions lasting for 45 minutes. Interventions will take place in facilities close to participants' work sites.

The financial feasibility of the effects of the interventions is calculated by using the Potential Model,[www.miljodata.se],which was created to calculate the financial feasibility of work health related measures. It differs from typical health economic cost-benefit analyses in the sense that it is aimed at simulating the economic consequences of an investment from a business point of view. In addition to the immediate real losses and sickness absences, the indirect financial consequences like effects on over time work are taken into account.

The rational of this study is to discover whether neuromuscular exercise and cognitive behavioral counseling are effective and economically feasible in reducing LBP and its' recurrence, and thus preventing chronic LBP, early retirement and disability pensions.

ELIGIBILITY:
Inclusion Criteria:

* woman aged 40 to 55
* working at one's current nursing job at least for 12 months
* intensity of LBP on Visual Analog Scale (VAS) has been greater than 20mm (scale 0-100) during the last month

Exclusion Criteria:

* serious former back injury (fracture, surgery, discus prolapse)
* chronic low back symptoms i.e. time when last experienced no low back pain is longer than six months
* pregnant or recent delivery (<12months)
* general health problems prevent moderate exercise
* body mass index >35

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 219 (Actual)
Dates: Start 2011-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Intensity of LBP for past month assessed by Visual Analog Scale | Baseline, 6, 12 and 24 months follow-up
  Changes in the intensity of LPB at the given time frame

SECONDARY OUTCOMES:
Movement control impairment | Baseline, 6, 12 and 24 months follow-up
  Changes in active movement control of the lower back will be assessed with six tests of movement control dysfunction introduced by Luomajoki et al.(2007, 2008, 2010). The test results have shown a significant difference between patients with LBP and healthy controls, as well as between patients with acute and chronic, and chronic and subacute LBP. Reliability of the tests has been established as well as responsiveness to physical exercise. For a subsample of participants the test performances will be videotaped to ensure the objectivity of the assessments.
Fear-avoidance beliefs questionnaire | Baseline, 6, 12 and 24 months follow-up
  Changes in fear-avoidance behaviour will be assed with the specific questionnaire on fear-avoidance beliefs (FABQ) addressing the behavior in both work and leisure (Waddel ym. 1993).
Objective assessment of physical activity with accelerometer | Baseline, 6, 12 and 24 months follow-up
  Objective assessment of physical activity is conducted at the given time points during seven consecutive days by accelerometers (Hookie AM 20 Activity Meter, Hookie Technologies Ltd, Espoo. Participants wear accelerometers at all times except for sleeping. Changes in physical activity patterns are investigated: total amount of sitting, light physical activity, moderate physical activity and strenuous physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Jaana H Suni, DSc, Docent, Principal Investigator — UKK Institute
Locations (1):
- UKK Institute for Health Promotion Reserach, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kolu P, Suni JH, Tokola K, Raitanen J, Rinne M, Taulaniemi A, Husu P, Kankaanpaa M, Parkkari J. Neuromuscular exercise and counseling for treating recurrent low back pain in female healthcare workers-Findings from a 24-month follow-up study of a randomized controlled trial. Scand J Med Sci Sports. 2023 Nov;33(11):2239-2249. doi: 10.1111/sms.14451. Epub 2023 Jul 19. PMID 37466018
- [Derived] Suni JH, Virkkunen T, Husu P, Tokola K, Parkkari J, Kankaanpaa M. Reliability and construct validity of the modified Finnish version of the 9-item patient health questionnaire and its associations within the biopsychosocial framework among female health-care workers with sub-acute or recurrent low back pain. BMC Musculoskelet Disord. 2021 Jan 7;22(1):37. doi: 10.1186/s12891-020-03832-y. PMID 33413235
- [Derived] Suni JH, Kolu P, Tokola K, Raitanen J, Rinne M, Taulaniemi A, Parkkari J, Kankaanpaa M. Effectiveness and cost-effectiveness of neuromuscular exercise and back care counseling in female healthcare workers with recurrent non-specific low back pain: a blinded four-arm randomized controlled trial. BMC Public Health. 2018 Dec 17;18(1):1376. doi: 10.1186/s12889-018-6293-9. PMID 30558592